CLINICAL TRIAL: NCT05084352
Title: Real Time Vital Sign Assessment to Predict Neurological Decline After Traumatic Brain Injury (RAPID-TBI)
Brief Title: Real Time Vital Sign Assessment to Predict Neurological Decline After Traumatic Brain Injury
Acronym: RAPID-TBI
Status: Recruiting | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Neeraj Badjatia, Professor, Department of Neurology, University of Maryland, Baltimore
Other Study IDs: HP-00087051
Record Dates: First submitted 2021-09-27; First posted 2021-10-19 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study will look to validate predictive algorithms developed in a previous study where we collected relevant data from trauma registry and after using advanced signal-processing and machine-learning, determined prediction scores regarding neuroworsening and other outcomes following traumatic brain injury.

ELIGIBILITY:
Inclusion Criteria:

* Arrival to the hospital within 6 hours of injury
* Age >= 18 years old
* Patients with traumatic brain injury(TBI). TBI is defined as any alteration or loss of consciousness with or without positive head C.T findings.

Exclusion Criteria:

* Deemed to have a non-survivable TBI
* Brain dead on arrival
* Active substance abuse for opiates and cocaine as noted by admission toxicology screen.
* Any thoracic or abdominal injury resulting in open surgical intervention
* Pregnancy
* Prisoners
* Active military
* Non - English speaking (due to necessity for consent in aims 2 and 3)
* Age > 89 years

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult TBI patients
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2021-03-29 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Neurological Decline | First 48 hours of injury
  Neurological decline is defined as a worsening in neurological status determined by a 2 point decline GCS, pupillary change, radiographic worsening defined by Rotterdam score, need for neurological or neurosurgical intervention (eg. treatment of seizure, raised ICP, hematoma evacuation)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided